CLINICAL TRIAL: NCT01771887
Title: Assessing the Effects of Education Program for Lebanese Diabetic Type 2 in Their Behavior of Auto Managing Their Sense of Self-efficacy and on Their Adhesion Therapy
Brief Title: Effects of Education Program for Lebanese Diabetic T2 in Their Behavior of Auto Managing, of Self-efficacy and Adhesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Randa Atallah, Ph.D. Candidate, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATALLAH-FSI-6
Record Dates: First submitted 2013-01-08; First posted 2013-01-18 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic Type2; education; self-management behaviors; self-efficacy; HbA1c
MeSH Terms: conditions — Diabetes Mellitus | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- education program (Experimental): education program in 6 hours for groups of 10 people. The content will be divided into 2 sessions with an interval of 2 weeks, the duration of each session is 3 hours. Means active learning, teaching materials in Arabic accompany the content masterful discussions on flipcharts, situation analysis, computer-assisted presentation, demonstration, 150 photos of Lebanese dishes. After, patients receive a 10-page illustrated book, a logbook of diabetes control. 2 weeks after the second education session, each participant will receive 5 calls every 15 days in 2 months. During each call, the research assistant will ask the patient about diet, exercise and self-monitoring, medication and foot care and this according to a checklist.
  Interventions: Behavioral: education program

INTERVENTIONS:
Behavioral: education program — education program in 6 hours and monitoring phone every 15 days

SUMMARY:
Diabetes mellitus is a disease of great frequency and is a major public health problem. In Lebanon, the incidence of diabetes is estimated at 12%, it is expected to double by the year 2025. Given the increasing prevalence of diabetes in Lebanon, the evolution of complications of this disease and the lack of studies at this level, it is appropriate to conduct a study that aims to evaluate the effects an education program for people with type 2 diabetes on their sense of self-efficacy and their ability to self-manage their disease to make them the most optimal therapeutic adherence possible. The design of this study is experimental type before / after randomization by diabetic patients. Education program delivered to the experimental group is the "Accu-Chek Education Program" of Roche. Membership will be assessed using a biomarker HbA1c should be <7%, and a questionnaire (Summary of Diabetes Self-Care Activities Measure), which measures self-care behaviors. Self-efficacy is measured using the Diabetes Management Self-Efficacy Scale. And this before the intervention and 3 months later. The sample will be 240 diabetic patients T2. Recruitment will be in outpatient diabetology a Hospital located in Beirut. Statistical analyzes used for descriptive variables are measures of central tendency, dispersion and frequency distribution. T-test and chi-square will be used to compare the socio-demographic characteristics of the 2 groups, experimental and control. To test hypotheses and determine the difference in the results of the dependent variables of the 2 groups, analysis of variance and covariance are used. The data will be processed using SPSS version 14.0.

DETAILED DESCRIPTION:
1. Following the implementation of a program of education, feeling of self-efficacy participants will be higher in the experimental group than in the control group.
2. Following the implementation of a program of education, self-management behaviors: monitoring the diet, the practice of physical exercise, self-monitoring blood sugar, taking medications and care feet, participants will be higher in the experimental group than in the control group.
3. Following the implementation of a program of education, the percentage of participants who have an HbA1c less than 7 will be higher in the experimental group than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Suffering from type 2 diabetes for at least one year,
* Lebanese speak, read and write Arabic,
* Have an HbA1c ≥ 7%

Exclusion Criteria:

* mental impairment
* a psychological problem uncontrolled and medicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
adhesion | HbA1c less than 7 % 3 months after the intervention

SECONDARY OUTCOMES:
Self-management behaviors | improvement of self-management behaviors 3 months after the intervention
  self-management behaviors will be measured using a questionnaire of 25 questions, Summary of Diabetes Self-Care Activities Measure SDSCA, which measures five behaviors: diet, exercise, self monitoring blood glucose, medication and foot care (Toobert et al., 2000).

OTHER OUTCOMES:
self-efficacy | enhancement of the sense of self-efficacy 3 months after the intervention
  Self-efficacy is measured using the Diabetes Management Self-Efficacy Scale (DMSES). This instrument was developed in 1999 by van der Bijl, van Poelgeest-Shortridge-Bagget & Eeltink. This instrument consists of 20 items.

CONTACTS AND LOCATIONS:
Overall Officials: José Côté, nur. Ph. D., Study Director — Université de Montréal
Locations (1):
- Outpatient of hospital of Hotel Dieu de France, Beirut, Lebanon